CLINICAL TRIAL: NCT01953419
Title: Pemetrexed for Previously Treated Patients With Metastatic Gastric Cancer: a Prospective Phase II Study
Brief Title: Phase II Study of Pemetrexed in Advanced or Recurrent Gastric Cancer After Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Vice president, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEM001
Record Dates: First submitted 2013-08-12; First posted 2013-10-01 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): received Pemetrexed disodium 500mg/m2 every 21 days until the presence of progressive disease or unacceptable toxicity
  Interventions: Drug: Pemetrexed disodium

INTERVENTIONS:
Drug: Pemetrexed disodium — Patients received Pemetrexed disodium 500mg/m2 every 21 days until the presence of progressive disease or unacceptable toxicity.Patients were instructed to take oral folic acid 400 mg daily beginning 5 days before the first therapy and until the final therapy. Patients received vitamin B12 before the first cycle of Pemetrexed and every three cycles of chemotherapy.
  Other Names: LY-231514; brand name: Alimta

SUMMARY:
This phase II trial aimed to assess the efficacy and safety of pemetrexed in patients with pretreated metastatic gastric cancer.

DETAILED DESCRIPTION:
Patients enrolled in this study received pemetrexed 500mg/m2, once every 21 days, until the presence of progressive disease or unacceptable toxicity. All patients took dexamethasone 3.75 mg twice daily, starting from the day before and continuing to the day after the drug administration. Patients were instructed to take oral folic acid 400 mg daily beginning 5 days before the first therapy and until the final therapy.Patients received Vitamin B12 very 3 cycle of chemoherapy. Granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF) or Erythropoietin (EPO) was not allowed, but they could be used when the patients suffered from bone marrow depression.

ELIGIBILITY:
Inclusion Criteria:

1. histological confirmed inoperable or metastatic adenocarcinoma of the stomach or gastro-esophageal junction
2. age between 18 and 80 years
3. ECOG performance status of 0 to 2
4. life expectancy ≥ 12 weeks
5. has measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST)
6. at least one prior chemotherapy regimen
7. adequate bone marrow function as defined by absolute neutrophil count more than or equal to 2000/mm3
8. platelet count more than or equal to 100,000/mm3 and hemoglobin more than or equal to 8 g/dL
9. adequate renal function defined by creatinine less than or equal to 1.25 × upper limit of normal(ULN) and creatinine clearance more than or equal to 60mL/min,
10. adequate liver function defined by bilirubin less than or equal to 1.0×ULN aspartate transferase(AST) and alanine transferase(ALT) less than or equal to 2.5 ×ULN.

Exclusion Criteria:

1. other primary malignancy
2. symptomatic central nervous system metastasis
3. pregnancy or lactation
4. cardiovascular events such as myocardial infarction in the previous 6 months or congestive heart failure
5. ongoing infection
6. inability or unwillingness to interrupt nonsteroidal anti-inflammatory drugs for 2 days before and after pemetrexed administration unwillingness to take folic acid or vitamin B12 supplementation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
ORR | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: RH Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen UniversityCancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No